CLINICAL TRIAL: NCT03285594
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, 52-week Multicenter Study to Evaluate the Efficacy and Safety of Sotagliflozin in Patients With Type 2 Diabetes Who Have Inadequate Glycemic Control on Basal Insulin Alone or in Addition to Oral Antidiabetes Drugs (OADs)
Brief Title: Efficacy and Safety of Sotagliflozin Versus Placebo in Participants With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control While Taking Insulin Alone or With Other Oral Antidiabetic Agents
Acronym: SOTA-INS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC14868; 2016-001804-43 (EudraCT Number); U1111-1190-7567 (Other: UTN)
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo (Placebo Comparator): Following a 4-week run-in period, participants were randomized to matching placebo to sotagliflozin 200 milligrams (mg) administered as 2 tablets, once daily, before the first meal of the day in the double-blind treatment period for up to 52 weeks. Background therapy with insulin glargine (with or without OADs) continued throughout the study.
  Interventions: Drug: Insulin glargine (HOE901); Drug: Placebo; Drug: Oral Antidiabetes Drugs (OADs)
- Sotagliflozin 200 mg (Experimental): Following a 4-week run-in period, participants were randomized to sotagliflozin 200 mg administered as 1 tablet and matching placebo as 1 tablet, once daily, before the first meal of the day in the double-blind treatment period for up to 52 weeks. Background therapy with insulin glargine (with or without OADs) continued throughout the study.
  Interventions: Drug: Sotagliflozin; Drug: Insulin glargine (HOE901); Drug: Placebo; Drug: Oral Antidiabetes Drugs (OADs)
- Sotagliflozin 400 mg (Experimental): Following a 4-week run-in period, participants were randomized to sotagliflozin 400 mg administered as 2 tablets, once daily, before the first meal of the day in the double-blind treatment period for up to 52 weeks. Background therapy with insulin glargine (with or without OADs) continued throughout the study.
  Interventions: Drug: Sotagliflozin; Drug: Insulin glargine (HOE901); Drug: Oral Antidiabetes Drugs (OADs)

INTERVENTIONS:
Drug: Sotagliflozin — Pharmaceutical form: Tablet
  Route of administration: Oral
  Other Names: SAR439954
  Arms: Sotagliflozin 200 mg; Sotagliflozin 400 mg
Drug: Insulin glargine (HOE901) — Pharmaceutical form: Solution
  Route of administration: Subcutaneous
  Other Names: Lantus
Drug: Placebo — Pharmaceutical form: Tablet
  Route of administration: Oral
  Arms: Placebo; Sotagliflozin 200 mg
Drug: Oral Antidiabetes Drugs (OADs) — OADs (including metformin) as prescribed by the investigator as per local labeling.

SUMMARY:
Primary Objective:

To demonstrate the superiority of sotagliflozin 400 milligrams (mg) versus placebo with respect to hemoglobin A1C (HbA1c) reduction in participants with type 2 diabetes mellitus (T2D) who have inadequate glycemic control on basal insulin alone or with oral antidiabetes drugs (OADs).

Secondary Objectives:

* To assess the effects of sotagliflozin 400 mg versus placebo on fasting plasma glucose (FPG), body weight, systolic blood pressure (SBP), and HbA1c.
* To assess the effects of sotagliflozin 200 mg versus placebo on HbA1c, body weight, FPG, and SBP.
* To evaluate the safety of sotagliflozin 400 and 200 mg versus placebo.

DETAILED DESCRIPTION:
Up to 60 weeks (Screening phase of up to 2 weeks, a 4-week Lantus titration/single-blind placebo Run-in phase), a 52-week double blind Treatment Period, and a 2-week post-treatment Follow-up Period.

ELIGIBILITY:
Inclusion criteria :

* Participants with Type 2 Diabetes Mellitus (T2DM) using any types of basal insulin alone or in combination with up to 2 OADs.
* Participants have given written informed consent to participate in the study in accordance with local regulations.

Exclusion criteria:

* At the time of Screening age <18 years or <legal age of majority, whichever is greater.
* Type 1 diabetes mellitus.
* Oral antidiabetic drugs dose not stable for 8 weeks before Screening.
* Use of basal insulin therapy (e.g., insulin glargine, Neutral Protamine Hagedorn (NPH), detemir, or degludec) for less than 6 months before Screening.
* Dose of basal insulin (e.g., insulin glargine, NPH, detemir, or degludec) not stable for 8 weeks before Screening (i.e., total daily insulin dose increased or decreased by more than 20%).
* Known unstable proliferative diabetic retinopathy or any other rapidly progressive diabetic retinopathy or macular edema that is likely to require laser, surgical treatment during study period.
* Use of injectable diabetes drugs other than basal insulin (e.g., insulin glargine, NPH, detemir, or degludec), i.e., prandial or rapid-acting insulins, short-acting insulins, glucagon-like peptide 1 (GLP-1) receptor agonists, or inhaled prandial insulin (Afrezza) within 8 weeks of Screening.
* Use of a selective sodium-glucose cotransporter type 2 (SGLT2) inhibitor (e.g., canagliflozin, dapagliflozin, or empagliflozin) within 3 months prior to the trial.
* Use of systemic glucocorticoids (excluding topical, intra articular, or ophthalmic application, nasal spray or inhaled forms) for more than 10 consecutive days within 90 days prior to the Screening Visit.
* Participants with severe anemia, severe cardiovascular (including congestive heart failure New York Heart Association IV), respiratory, hepatic, neurological, psychiatric, or active malignant tumor or other major systemic disease that, according to the Investigator, will preclude their safe participation in this study, or will make implementation of the protocol or interpretation of the study results difficult.
* Lower extremity complications (such as skin ulcers, infection, osteomyelitis and gangrene) identified during the Screening period, and still requiring treatment at Randomization.
* Known presence of factors that interfere with the Central Lab HbA1c measurement (e.g., genetic hemoglobin (Hb) variants) compromising the reliability of HbA1c assessment or medical conditions that affect interpretation of HbA1c results (e.g., blood transfusion or severe blood loss in the last 3 months prior to randomization, any condition that shortens erythrocyte survival).
* Participants who has taken other investigational drugs or prohibited therapy for this study within 12 weeks or 5 half-lives from prior to Screening, whichever is longer.
* Participants unwilling to perform self-monitoring of blood glucose (SMBG), complete the patient diary, or comply with study visits and other study procedures as required per protocol.
* HbA1c <7.5% or HbA1c >10.5% measured by the central laboratory at Screening.
* HbA1c <7% measured by the central laboratory at Visit 5 (Week -1).
* History of diabetic ketoacidosis or nonketotic hyperosmolar coma within 12 weeks prior to the Screening Visit.
* Pregnant (confirmed by serum pregnancy test at Screening) or breastfeeding women.
* Women of childbearing potential not willing to use highly effective method(s) of birth control during the study treatment period and the follow-up period, or who are unwilling or unable to be tested for pregnancy during the study.
* Mean of 3 separate blood pressure measurements >180 mmHg (systolic blood pressure [SBP]) or >100 mmHg (diastolic blood pressure [DBP]).
* History of gastric surgery including history of gastric banding or inflammatory bowel disease within 3 years prior to the Screening Visit.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 times the upper limit of the normal laboratory range
* Total bilirubin >1.5 times the upper limit of the normal laboratory range (except in case of Gilbert's syndrome).

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suman Wason, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (106):
- United States (50):
  - Investigational Site Number 8406028, Mesa, Arizona
  - Investigational Site Number 8406013, Phoenix, Arizona
  - Investigational Site Number 8406020, Phoenix, Arizona
  - Investigational Site Number 8406006, Huntington Park, California
  - Investigational Site Number 8406053, Lincoln, California
  - Investigational Site Number 8406040, Los Angeles, California
  - Investigational Site Number 8406043, Coral Gables, Florida
  - Investigational Site Number 8406008, DeLand, Florida
  - Investigational Site Number 8406030, Maitland, Florida
  - Investigational Site Number 8406003, New Port Richey, Florida
  - Investigational Site Number 8406029, North Miami Beach, Florida
  - Investigational Site Number 8406052, Ocoee, Florida
  - Investigational Site Number 8406001, Port Charlotte, Florida
  - Investigational Site Number 8406022, St. Petersburg, Florida
  - Investigational Site Number 8406025, Tampa, Florida
  - Investigational Site Number 8406002, West Palm Beach, Florida
  - Investigational Site Number 8406054, Chicago, Illinois
  - Investigational Site Number 8406027, Chicago, Illinois
  - Investigational Site Number 8406042, Evansville, Indiana
  - Investigational Site Number 8406044, New Orleans, Louisiana
  - Investigational Site Number 8406051, New Orleans, Louisiana
  - Investigational Site Number 8406024, Rockville, Maryland
  - Investigational Site Number 8406016, Detroit, Michigan
  - Investigational Site Number 8406011, St Louis, Missouri
  - Investigational Site Number 8406010, Papillion, Nebraska
  - Investigational Site Number 8406018, New York, New York
  - Investigational Site Number 8406034, Asheville, North Carolina
  - Investigational Site Number 8406046, Chapel Hill, North Carolina
  - Investigational Site Number 8406026, Charlotte, North Carolina
  - Investigational Site Number 8406038, Greenville, North Carolina
  - Investigational Site Number 8406036, Hickory, North Carolina
  - Investigational Site Number 8406015, Wilmington, North Carolina
  - Investigational Site Number 8406019, Winston-Salem, North Carolina
  - Investigational Site Number 8406031, Beachwood, Ohio
  - Investigational Site Number 8406023, Columbus, Ohio
  - Investigational Site Number 8406005, Dublin, Ohio
  - Investigational Site Number 8406004, Mentor, Ohio
  - Investigational Site Number 8406033, Oklahoma City, Oklahoma
  - Investigational Site Number 8406032, Moncks Corner, South Carolina
  - Investigational Site Number 8406009, Chattanooga, Tennessee
  - Investigational Site Number 8406045, Seymour, Tennessee
  - Investigational Site Number 8406047, Dallas, Texas
  - Investigational Site Number 8406017, Dallas, Texas
  - Investigational Site Number 8406048, Houston, Texas
  - Investigational Site Number 8406037, Houston, Texas
  - Investigational Site Number 8406039, McAllen, Texas
  - Investigational Site Number 8406050, San Antonio, Texas
  - Investigational Site Number 8406021, Shavano Park, Texas
  - Investigational Site Number 8406035, Salt Lake City, Utah
  - Investigational Site Number 8406014, West Jordan, Utah
- Bulgaria (9):
  - Investigational Site Number 1006009, Gabrovo
  - Investigational Site Number 1006003, Plovdiv
  - Investigational Site Number 1006004, Rousse
  - Investigational Site Number 1006001, Rousse
  - Investigational Site Number 1006006, Smolyan
  - Investigational Site Number 1006002, Sofia
  - Investigational Site Number 1006010, Sofia
  - Investigational Site Number 1006005, Stara Zagora
  - Investigational Site Number 1006007, Varna
- Canada (5):
  - Investigational Site Number 1246003, Brampton
  - Investigational Site Number 1246005, Burlington
  - Investigational Site Number 1246004, Etobicoke
  - Investigational Site Number 1246002, Toronto
  - Investigational Site Number 1246001, Vancouver
- Czechia (7):
  - Investigational Site Number 2036003, Holešov
  - Investigational Site Number 2036002, Krnov
  - Investigational Site Number 2036001, Olomouc
  - Investigational Site Number 2036005, Ostrava
  - Investigational Site Number 2036007, Prague
  - Investigational Site Number 2036008, Prague
  - Investigational Site Number 2036006, Praha 10 - Uhrineves
- France (11):
  - Investigational Site Number 2506008, Besançon
  - Investigational Site Number 2506003, Corbeil-Essonnes
  - Investigational Site Number 2506005, Dijon
  - Investigational Site Number 2506012, Mulhouse
  - Investigational Site Number 2506004, Nantes
  - Investigational Site Number 2506007, Narbonne
  - Investigational Site Number 2506006, Paris
  - Investigational Site Number 2506010, Pierre-Bénite
  - Investigational Site Number 2506009, Poitiers
  - Investigational Site Number 2506011, Saint-Mandé
  - Investigational Site Number 2506002, Vénissieux
- Hungary (8):
  - Investigational Site Number 3486007, Budapest
  - Investigational Site Number 3486002, Budapest
  - Investigational Site Number 3486006, Hatvan
  - Investigational Site Number 3486009, Kecskemét
  - Investigational Site Number 3486003, Komárom
  - Investigational Site Number 3486005, Nyíregyháza
  - Investigational Site Number 3486001, Pécs
  - Investigational Site Number 3486008, Zalaegerszeg
- Slovakia (10):
  - Investigational Site Number 7036004, Bardejov
  - Investigational Site Number 7036008, Bratislava
  - Investigational Site Number 7036001, Bratislava
  - Investigational Site Number 7036010, Košice
  - Investigational Site Number 7036003, Košice
  - Investigational Site Number 7036007, Levice
  - Investigational Site Number 7036009, Levice
  - Investigational Site Number 7036011, Lučenec
  - Investigational Site Number 7036006, Nitra
  - Investigational Site Number 7036005, Sabinov
- United Kingdom (6):
  - Investigational Site Number 8266002, Darlington
  - Investigational Site Number 8266006, Doncaster
  - Investigational Site Number 8266008, Dundee
  - Investigational Site Number 8266001, Leicester
  - Investigational Site Number 8266004, London
  - Investigational Site Number 8266003, Salford

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 101 investigative sites in the United States, Bulgaria, Canada, Czech Republic, France, Hungary, Slovakia, the United Kingdom from 15 September 2017 to 27 September 2019.
Pre-assignment Details: Participants with a diagnosis of Type 2 Diabetes Mellitus were enrolled in 1 of 3 treatment groups, placebo, sotagliflozin 200 milligrams (mg) and sotagliflozin 400 mg. Participants were randomized at a ratio of 1:1:2 respectively to 1 of 3 groups.
Groups:
- Placebo: Following a 4-week run-in period, participants were randomized to receive matching placebo to sotagliflozin 200 mg administered as 2 tablets, once daily, before the first meal of the day in the double-blind treatment period for up to 55.7 weeks. Background therapy with insulin glargine (with or without oral antidiabetes drugs [OADs]) continued throughout the study.
- Sotagliflozin 200 mg: Following a 4-week run-in period, participants were randomized to sotagliflozin 200 mg administered as 1 tablet and matching placebo as 1 tablet, once daily, before the first meal of the day in the double-blind treatment period for up to 54.7 weeks. Background therapy with insulin glargine (with or without OADs) continued throughout the study.
- Sotagliflozin 400 mg: Following a 4-week run-in period, participants were randomized to sotagliflozin 400 mg administered as 2 tablets, once daily, before the first meal of the day in the double-blind treatment period for up to 54.6 weeks. Background therapy with insulin glargine (with or without OADs) continued throughout the study.
Period: Overall Study
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Started | 144 | 141 | 286
Treated | 144 | 141 | 285
Completed | 129 | 130 | 249
Not Completed | 15 | 11 | 37
Not completed — At the Participant's Own Request | 10 | 5 | 21
Not completed — Adverse Event | 2 | 2 | 6
Not completed — Poor Compliance to Protocol | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Reason Not Specified | 3 | 4 | 8

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants irrespective of compliance with the study protocol and procedures.
Groups:
- Placebo: Following a 4-week run-in period, participants were randomized to receive matching placebo to sotagliflozin 200 mg administered as 2 tablets, once daily, before the first meal of the day in the double-blind treatment period for up to 55.7 weeks. Background therapy with insulin glargine (with or without OADs) continued throughout the study.
- Total: Total of all reporting groups
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg | Total
Number analyzed (Participants) | 144 | 141 | 286 | 571
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (8.9) | 62.1 (10.2) | 62.7 (9.1) | 62.4 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 65 | 132 | 255
  Male | 86 | 76 | 154 | 316
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 25 | 42 | 79
  Not Hispanic or Latino | 129 | 113 | 239 | 481
  Unknown or Not Reported | 3 | 3 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 2 | 5
  Asian | 9 | 1 | 6 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 3 | 3
  Black or African American | 10 | 10 | 27 | 47
  White | 117 | 124 | 234 | 475
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 5 | 5 | 13 | 23
Region of Enrollment [Number; unit: participants]
  Bulgaria | 9 | 13 | 35 | 57
  Canada | 7 | 6 | 16 | 29
  Czechia | 14 | 11 | 24 | 49
  France | 8 | 8 | 14 | 30
  Hungary | 12 | 13 | 21 | 46
  Slovakia | 24 | 21 | 32 | 77
  United Kingdom | 0 | 0 | 4 | 4
  United States | 70 | 69 | 140 | 279
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percentage of HbA1c] | 8.76 (0.79) | 8.76 (0.83) | 8.69 (0.80) | 8.72 (0.80)
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: millimeter of Mercury (mmHg)] | 137.59 (14.12) | 136.40 (15.54) | 135.84 (14.95) | 136.42 (14.89)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at Week 18
Description: An analysis of covariance (ANCOVA) model was used for the analysis.
Time Frame: Baseline and Week 18
Population: Intent-to-treat (ITT) population included all randomized participants irrespective of compliance with the study protocol and procedures. Missing data are imputed using washout multiple imputation method under the missing not at random framework.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 144 | 141 | 286
percentage of HbA1c | -0.27 (0.073) | -0.72 (0.073) | -0.81 (0.056)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; The change from baseline to Week 18 was analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at Week -1, randomization strata of mean SBP (<130, ≥130 mmHg) at Week -1, randomization strata of sulfonylureas use (yes, no) at Week -1, and country as fixed effects, and baseline HbA1c as a covariate; Test type: Superiority; p < 0.0001, ANCOVA; Difference in Least Square (LS) Means = -0.45, 95% CI 2-sided [-0.638 to -0.271], Standard Error of Mean 0.094
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LS Means = -0.55, 95% CI 2-sided [-0.706 to -0.387], Standard Error of Mean 0.081

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 18
Description: FPG was performed in fasting state, that is, without any food intake (except for water) for at least 8 hours. An ANCOVA model was used for the analysis.
Time Frame: Baseline and Week 18
Population: ITT population included all randomized participants irrespective of compliance with the study protocol and procedures. Missing data are imputed using washout multiple imputation method under the missing not at random framework.
Measure: Least Squares Mean (Standard Error); unit: milligram per deciliter (mg/dL)
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 144 | 141 | 286
milligram per deciliter (mg/dL) | 12.882 (3.6045) | -2.975 (3.6083) | -8.949 (2.7550)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; The change from baseline to Week 18 was analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at Week -1, randomization strata of mean SBP (<130, ≥130 mmHg) at Week -1, randomization strata of sulfonylureas use (yes, no) at Week -1, and country as fixed effects, and baseline FPG as a covariate; Test type: Superiority; p = 0.0006, ANCOVA; Difference in LS Means = -15.858, 95% CI 2-sided [-24.8845 to -6.8309], Standard Error of Mean 4.6056
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LS Means = -21.832, 95% CI 2-sided [-29.7725 to -13.8911], Standard Error of Mean 4.0514

3. Secondary Outcome: Change From Baseline in Body Weight at Week 18
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline and Week 18
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 144 | 141 | 286
kilogram (kg) | 0.36 (0.249) | -0.73 (0.250) | -1.37 (0.190)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; The change from baseline to Week 18 is analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at Week -1, randomization strata of mean SBP (<130, ≥130 mmHg) at Week -1, randomization strata of sulfonylureas use (yes, no) at Week -1, and country as fixed effects, and baseline body weight as a covariate; Test type: Superiority; p = 0.0007, ANCOVA; Difference in LS Means = -1.09, 95% CI 2-sided [-1.716 to -0.462], Standard Error of Mean 0.32
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LS Means = -1.73, 95% CI 2-sided [-2.274 to -1.183], Standard Error of Mean 0.278

4. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) for Participants With Baseline SBP ≥130 mmHg at Week 12
Description: An ANCOVA model was used for the analysis. Here, N is the number of participants with data available at a given time point.
Time Frame: Baseline and Week 12
Population: Analysis population included participants with baseline SBP ≥ 130 mmHg in ITT population where, ITT population included all randomized participants irrespective of compliance with the study protocol and procedures. Missing data are imputed using washout multiple imputation method under the missing not at random framework.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 88 | 92 | 171
mmHg | -4.67 (1.470) | -8.58 (1.447) | -8.50 (1.103)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; The change from baseline to Week 12 was analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at Week -1, randomization strata of sulfonylureas use (yes, no) at Week -1, and country as fixed effects, and baseline SBP as a covariate; Test type: Superiority; p = 0.04, ANCOVA; Difference in LS Means = -3.91, 95% CI 2-sided [-7.642 to -0.178], Standard Error of Mean 1.904
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0239, ANCOVA; Difference in LS Means = -3.83, 95% CI 2-sided [-7.161 to -0.507], Standard Error of Mean 1.697

5. Secondary Outcome: Change From Baseline in SBP at Week 12 for All Participants
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 144 | 141 | 286
mmHg | -0.21 (1.120) | -5.15 (1.117) | -4.10 (0.867)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; The change from baseline to Week 12 was analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at Week -1, randomization strata of mean SBP (<130, ≥130 mmHg) at Week -1, randomization strata of sulfonylureas use (yes, no) at Week -1, and country as fixed effects, and baseline SBP as a covariate; Test type: Superiority; Difference in LS Means = -4.94, 95% CI 2-sided [-7.73 to -2.142], Standard Error of Mean 1.425
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0018, ANCOVA; Difference in LS Means = -3.89, 95% CI 2-sided [-6.333 to -1.448], Standard Error of Mean 1.246

6. Secondary Outcome: Change From Baseline in HbA1c at Week 52
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline and Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 144 | 141 | 286
percentage of HbA1c | 0.00 (0.279) | -0.52 (0.152) | -0.57 (0.114)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; The change from baseline to Week 52 was analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at Week -1, randomization strata of mean SBP (<130, ≥130 mmHg) at Week -1, randomization strata of sulfonylureas use (yes, no) at Week -1, and country as fixed effects, and baseline HbA1c as a covariate; Test type: Superiority; p = 0.1265, ANCOVA; Difference in LS Means = -0.52, 95% CI 2-sided [-1.185 to 0.147], Standard Error of Mean 0.34
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.074, ANCOVA; Difference in LS Means = -0.57, 95% CI 2-sided [-1.199 to 0.055], Standard Error of Mean 0.32

7. Secondary Outcome: Change From Baseline in Body Weight at Week 52
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline and Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 144 | 141 | 286
kg | -0.18 (0.579) | -1.19 (0.620) | -0.83 (0.374)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; The change from baseline to Week 18 was analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at Week -1, randomization strata of mean SBP (<130, ≥130 mmHg) at Week -1, randomization strata of sulfonylureas use (yes, no) at Week -1, and country as fixed effects, and baseline body weight as a covariate; Test type: Superiority; p = 0.2466, ANCOVA; Difference in LS Means = -1.01, 95% CI 2-sided [-2.707 to 0.696], Standard Error of Mean 0.868
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.332, ANCOVA; Difference in LS Means = -0.65, 95% CI 2-sided [-1.969 to 0.665], Standard Error of Mean 0.672

8. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participants or clinical investigation participants administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: First dose of study drug to last dose of study drug (up to 55.7 weeks) + 2 weeks
Population: Safety population included all randomized participants who received at least 1 dose of double-blind investigational medicinal product (IMP) (regardless of the amount of treatment administered).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 144 | 141 | 285
percentage of participants | 64.6 | 54.6 | 59.3

9. Other Pre Specified Outcome: Percentage of Participants With Hypoglycemic Events
Description: Percentage of participants with hypoglycemic events are reported for the following 3 categories: Any hypoglycemia (as reported in the Electronic Case Report Form); Documented symptomatic hypoglycemia [typical symptoms of hypoglycemia (increased sweating, nervousness, asthenia/weakness, tremor, dizziness, increased appetite, palpitations, headache, sleep disorder, confusion, seizures, unconsciousness, and/or coma) and plasma glucose ≤ 70 mg/dL (3.9 mmol/L)]; Severe [an event requiring assistance of another person to actively administer carbohydrate, glucagon, intravenous glucose or other resuscitative actions] or documented symptomatic hypoglycemia [typical symptoms of hypoglycemia and plasma glucose ≤ 70 mg/dL].
Time Frame: Up to 55.7 weeks
Population: Safety population included all randomised participants who received at least 1 dose of double-blind investigational medicinal product (IMP) (regardless of the amount of treatment administered).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 144 | 141 | 285
percentage of participants
  Any hypoglycemia | 62.5 | 56.0 | 62.8
  Documented symptomatic hypoglycemia | 44.4 | 41.8 | 46
  Severe or documented symptomatic hypoglycemia | 44.4 | 41.8 | 46

ADVERSE EVENTS:
Time Frame: Deaths: Up to approximately 60 weeks; Adverse Events: First dose of study drug to last dose of study drug (up to 55.7 weeks) + 2 weeks
Description: Safety population included all randomized participants who had received at least 1 dose of double-blind investigational medicinal product (regardless of the amount of treatment administered). Hypoglycemia was captured and handled separately from other adverse events and is reported in the outcome measure section.
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
All-Cause Mortality (participants affected / at risk) | 2/144 | 1/141 | 6/285
Serious Adverse Events (participants affected / at risk) | 16/144 | 19/141 | 28/285
Other Adverse Events (participants affected / at risk) | 30/144 | 18/141 | 45/285
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=144) | Sotagliflozin 200 mg (N=141) | Sotagliflozin 400 mg (N=285)
Aortic stenosis (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Sudden cardiac death (General disorders) | 1 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 1
Postoperative thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | 2
Angina unstable (Cardiac disorders) | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Reperfusion arrhythmia (Cardiac disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0 | 0
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Retinal artery thrombosis (Eye disorders) | 0 | 0 | 1
Retinopathy proliferative (Eye disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Renal haematoma (Renal and urinary disorders) | 0 | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 1
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Infected bite (Infections and infestations) | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0 | 1
Osteomyelitis acute (Infections and infestations) | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Pyelonephritis chronic (Infections and infestations) | 0 | 0 | 1
Renal abscess (Infections and infestations) | 0 | 1 | 0
Scrotal abscess (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Enlarged uvula (Gastrointestinal disorders) | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=144) | Sotagliflozin 200 mg (N=141) | Sotagliflozin 400 mg (N=285)
Vitamin D deficiency (Metabolism and nutrition disorders) | 9 | 4 | 10
Nasopharyngitis (Infections and infestations) | 7 | 9 | 14
Upper respiratory tract infection (Infections and infestations) | 8 | 1 | 14
Urinary tract infection (Infections and infestations) | 8 | 6 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution must provide any proposed publication or presentation to Sponsor for Sponsor's review, comment and approval at least thirty (30) days prior to the proposed submission for publication date or the proposed presentation date. Sponsor shall have the right to have deleted from the final version of the publication any confidential information, proprietary information, or patentable subject matter.

DOCUMENTS (2):
  • Study Protocol (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/94/NCT03285594/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/94/NCT03285594/SAP_001.pdf